CLINICAL TRIAL: NCT06290869
Title: Providing Tobacco Treatment to Patients Undergoing Lung Cancer Screening at MedStar Health: A Randomized Trial (Tobacco Education and Lung Health Study)
Brief Title: Tobacco Education and Lung Health Study (TEAL)
Acronym: TEAL
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Principal Investigator, Kathryn L. Taylor, Ph.D., Professor, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00006070
Record Dates: First submitted 2024-02-15; First posted 2024-03-04 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Smoking Cessation
Keywords: high risk for lung cancer
MeSH Terms: conditions — Smoking Cessation | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MedStar Health System (Experimental): Phone-based Tobacco Treatment, Nicotine Replacement, and Stepped Care Intervention
  Interventions: Behavioral: Phone-based Tobacco Treatment, Nicotine Replacement, and Stepped Care Intervention
- E-Referral to the Tobacco Quitline (Active Comparator): Standard tobacco quitline protocol, including coaching, nicotine replacement, and web-, and text-based resources.
  Interventions: Behavioral: E-Referral to the Tobacco Quitline

INTERVENTIONS:
Behavioral: Phone-based Tobacco Treatment, Nicotine Replacement, and Stepped Care Intervention — In the MedStar Health System (MHS) arm, we offer 5 phone sessions with a tobacco treatment specialist (TTS) during the first 3 months of treatment plus combination nicotine replacement (patches and lozenges). For those who have not quit at 3 months, 50% will be randomly assigned to stepped care (3 phone sessions with RN/NP + prescription medications as needed) vs. the continued TTS + NRT intervention. Those who have quit at 3 months will be offered 3 relapse prevention phone sessions with the TTS. Thus, all are offered 8 sessions. The TTS will use motivational interviewing to address ambivalence about quitting, education about the risks of continued smoking, encouragement to use and adhere to NRT, and the impact of the screening result (the teachable moment) by framing it as a potential motivator or opportunity to reduce future health risks and to maximize quality of life.
  Arms: MedStar Health System
Behavioral: E-Referral to the Tobacco Quitline — In the Quitline E-Referral arm, an e-referral will be generated from the EHR by our staff, will be signed by the LCS ordering provider and sent to the quitline through the closed-looped quitline's success.58-61,123 The quitline is an important comparator, given that it is an evidence-based and low-cost intervention already employed by many LCS sites system and the standard quitline protocol will then occur: 5 proactive contact attempts, up to 5 sessions, and up to 8 weeks of free NRT (depending on supplies). Quitline counselors are highly trained to conduct cessation treatment and extensive research has validated the quitline's success. The quitline is an important comparator, given that it is an evidence-based and low-cost intervention already employed by many LCS sites.
  Arms: E-Referral to the Tobacco Quitline

SUMMARY:
Primary Objective To compare two smoking cessation interventions among individuals undergoing lung cancer screening. Primary outcomes are: 3-month self-reported abstinence from cigarettes and 6-month self-reported and bioverified abstinence from cigarettes.

Secondary Objectives 1) To evaluate reach and engagement overall and by subgroup (e.g., race and ethnicity, underinsured, readiness to quit). 2) To conduct an economic analysis to evaluate intervention costs from the health system perspective.

DETAILED DESCRIPTION:
Providing smoking cessation treatment in conjunction with the recently expanded lung cancer screening guidelines is estimated to substantially reduce lung cancer deaths and increase life-years gained compared to conducting lung screening alone. Although CMS recommends that individuals undergoing lung screening who currently smoke are offered cessation treatment, there are multiple barriers to treatment delivery. Improving the evidence-base of cessation treatment for patients undergoing lung screening and methods to promote the systematic uptake of cessation treatment into routine practice, particularly among diverse populations, is essential for realizing the maximum benefit of lung screening. Guided by the Practical, Robust, Implementation & Sustainability framework, we will extend our prior work (CA R01207228). We propose a health system-level, pragmatic, randomized trial to compare the effectiveness of two evidence-based cessation treatments, with implementation strategies designed to address barriers to reach and engagement, particularly among underserved groups (e.g., racial and ethnic minority groups, underinsured patients, and patients not ready to quit) who are less likely to receive cessation treatment. To maximize generalizability to other health systems and to improve reach among heterogeneous groups, all patients scheduled at one of the 10 lung screening sites at MedStar Health, the largest and most diverse health system in the Mid-Atlantic, will be identified via the EHR, contacted for enrollment using an opt-out approach, and randomized to: 1) Quitline E-referral (QL-E; N=594) via the EHR and quitline integrated system, including proactive outreach and standard phone-based counseling + nicotine replacement provided by the quitline vs. 2) MedStar Health System (MHS; N=594), centralized, phone-based + NRT intervention adapted and improved from our prior trial, with a randomized stepped care intervention for those who are not abstinent at 3 months. Specific aims are: 1. To compare e-referral to the Quitline vs. the centralized Health System intervention. Primary outcomes are: 3-month self-reported abstinence from cigarettes and 6-month self-reported and bioverified abstinence from cigarettes. We will assess intervention mediators (e.g., treatment engagement) and moderators (e.g., readiness to quit) at 6-months. 2. To evaluate reach and engagement overall and by subgroup (e.g., race and ethnicity, underinsured, readiness to quit) and using mixed-methods to understand the contextual factors related to the feasibility and acceptability of the interventions and implementation strategies. 3. To conduct an economic analysis to evaluate costs, average and incremental cost per quit, and budget impact of the intervention at 3- and 6-months from the health system p0erspective. Proposal strengths include testing the effectiveness and economic outcomes of two cessation interventions while simultaneously laying the groundwork for future implementation within this and other diverse health systems. Our innovative approach capitalizes on the EHR for recruitment, provides multilevel training focused on diverse populations, and accounts for intervention context to inform future care delivery.

ELIGIBILITY:
Inclusion Criteria:

* eligible for a screening or diagnostic scan,
* USPSTF eligibility criteria (50-80 years old and >20-pack years);
* currently smoking cigarettes (>1 in the past 30 days);
* English speaking;
* able to provide meaningful consent.

Exclusion Criteria:

* prior lung cancer,
* hearing impairment,
* cognitive impairment,
* household member already enrolled.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1188 (Estimated)
Dates: Start 2024-02-22 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Biochemically verified smoking abstinence- MHS vs. QL-E arms | 6-month assessment
  Biochemically verified 7-day point prevalence abstinence rates, comparing the Health System (MHS) arm and the Quitline (QL-E) arm
Biochemically verified smoking abstinence--continued MHS arm vs Stepped Care | 6-month assessment
  Biochemically verified 7-day abstinence rates between the Stepped Care arm and the Continued MHS arm

SECONDARY OUTCOMES:
self-reported smoking status | 3-month and 6-month assessments
  self-reported abstinence (defined as in the past 7 days and in the past 30 days)
cigarettes per day | 3-month and 6-month assessments
  number of cigarettes smoked per day
readiness to quit | 3-month and 6-month assessments
  readiness to quit (defined as ready to quit in the next 30 days, the next six months, or not ready to quit)
Patient reach and patient engagement | Assessed through study completion, an average of six months.
  Reach: % of eligible smokers enrolled in trial; Engagement: % who receive the intervention, both overall and among subgroups
Costs per arm from the health system perspective | Assessed through study completion, an average of six months.
  Staff time costs; fixed costs, and variable costs

CONTACTS AND LOCATIONS:
Locations (1):
- Georgetown University Medical Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes